CLINICAL TRIAL: NCT00863512
Title: A Randomized Phase III Trial of Adjuvant Chemotherapy in Patients With Early Stage Non-Small Cell Lung Cancer Associated With Banking of Frozen Tumor Specimens and Collection of Gene Expression Profile Data
Brief Title: Chemotherapy or Observation in Treating Patients With Early Stage Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30506; CALGB-30506; CDR0000636895 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Cisplatin; Docetaxel; Gemcitabine; Pemetrexed; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive cisplatin IV on day 1 and vinorelbine ditartrate IV on days 1 and 8 OR docetaxel IV and cytarabine IV on day 1 OR gemcitabine hydrochloride IV on days 1 and 8 and cytarabine IV on day 1 OR pemetrexed disodium IV and cisplatin IV on day 1.. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium; Drug: vinorelbine tartrate
- Arm II (Experimental): Patients receive standard care (observation).
  Interventions: Procedure: standard follow-up care

INTERVENTIONS:
Drug: cisplatin — Given IV
  Arms: Arm I
Drug: docetaxel — Given IV
  Arms: Arm I
Drug: gemcitabine hydrochloride — Given IV
  Arms: Arm I
Drug: pemetrexed disodium — Given IV
  Arms: Arm I
Drug: vinorelbine tartrate — Given IV
  Arms: Arm I
Procedure: standard follow-up care — Standard care
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinorelbine, cisplatin, docetaxel, gemcitabine, and pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sometimes after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether chemotherapy is more effective than observation in treating patients who have undergone surgery for stage I non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying four chemotherapy regimens to see how well they work compared with observation in treating patients with early stage non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the potential overall survival benefit of adjuvant chemotherapy in patients with early stage non-small cell lung cancer (NSCLC) randomized to chemotherapy compared to those randomized to the present standard of care (observation).
* To collect and process high-quality fresh frozen lung cancer tumor tissue for gene expression array generation from multiple institutions.

Secondary

* To evaluate selected genomic-based lung cancer prognostic models using data from the patients randomized to observation after resection.
* To characterize the rate of chemotherapy toxicity for the different chemotherapy treatment regimens.
* To assess quality of life (QOL) in early stage patients periodically after resection for NSCLC.
* To examine the impact of chemotherapy on QOL for patients receiving chemotherapy, as compared to patients in the observation arm.

OUTLINE: This is a multicenter study. Patients are stratified according to pathologic stage (I vs II) and ECOG performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms within 12 weeks after surgery.

All patients undergo complete resection of disease (i.e., lobectomy, sleeve lobectomy, bi-lobectomy, or pneumonectomy, but not segmentectomy or wedge resection).

* Arm I: Patients receive 1 of 3 chemotherapy regimens. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

  * Regimen 1: Patients receive vinorelbine ditartrate IV over 10 minutes on days 1 and 8 and cisplatin IV over 60 minutes on day 1.
  * Regimen 2: Patients receive docetaxel IV over 60 minutes and cisplatin IV over 60 minutes on day 1.
  * Regimen 3: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 60 minutes on day 1.
  * Regimen 4: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 60 minutes on day 1.
* Arm II: Patients receive standard care (observation). Tissue obtained at surgery is examined by RNA microarray analysis. A Lung Metagene Score (LMS) is determined for each patient and correlated with survival and response.

After completion of study treatment, patients are followed every 6 months for 5 years and then once a year for 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Any variant allowed (e.g., pure or mixed bronchioloalveolar carcinoma or adenosquamous cell carcinoma)
  * Primary tumor must be T1a, T1b, T2a, or T2b by AJCC 7.0
  * No status
* Tumor measuring ≥ 2.0 cm but ≤ 7.0 cm in diameter by CT scan

  * The mass must have a source document to verify tumor size in the greatest dimension, which includes a CT scan report, a clinic note from the enrolling physician, and/or a printed image with caliper measurements on the lung mass
* Node-negative disease

  * Evidence of hilar or mediastinal node involvement by chest CT scan (> 1 cm diameter) must be assessed with mediastinoscopy, endo-esophageal ultrasound with biopsy, endo-bronchial ultrasound, bronchoscopy, or mediastinal nodal sampling before or at time of thoracotomy
* No locally advanced or metastatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Granulocytes ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Bilirubin ≤ 1.5 mg/dL
* AST < 1.5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of prior or concurrent malignancy, except curatively treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, surgically treated in situ carcinoma of the breast, or other cancer for which the patient has been disease-free for 3 years

PRIOR CONCURRENT THERAPY:

* More than 3 years since prior cytotoxic or anticancer treatment
* No concurrent treatment with hormones or other chemotherapeutic agents, except steroids given for adrenal failure, hormone administered for nondisease-related conditions (e.g., insulin for diabetes), or intermittent use of dexamethasone as an antiemetic
* No concurrent thoracic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Harpole, MD, Study Chair — Duke Cancer Institute
Locations (94):
- United States (93):
  - Regional Medical Center, Anniston, Alabama
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Pismo Beach, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Saint Francis Hospital Cancer Center, Poughkeepsie, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
- St. Vincent's Hospital - Melbourne, Fitzroy, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Chemotherapy): Patients receive cisplatin 75 mg/m^2 by IV on day 1 and vinorelbine ditartrate 30 mg/m^2 by IV on days 1 and 8 OR docetaxel 75 mg/m^2 by IV and cisplatin 75 mg/m^2 by IV on day 1 OR gemcitabine hydrochloride 1200 mg/m^2 by IV on days 1 and 8 and cisplatin 75 mg/m^2 by IV on day 1 OR pemetrexed disodium 500 mg/m^2 by IV and 75 mg/m^2 by cisplatin IV on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm II (Observation): Patients receive standard care (observation).
Period: Overall Study
Arm/Group | Arm I (Chemotherapy) | Arm II (Observation)
Started | 17 | 17
Completed | 3 | 17
Not Completed | 14 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 11 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy) | Arm II (Observation) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Full Range); unit: years] | 67 [43 to 78] | 63 [49 to 77] | 67 [43 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 1 | 3
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time between formal registration and death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Up to 12 years
Population: Study terminated prematurely with 34 participants recruited. Per protocol, 338 events were needed to conduct the primary analysis; therefore, the planned analyses was not performed due to a lack of events and a termination of data collection.
Arm/Group | Arm I (Chemotherapy) | Arm II (Observation)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Data is available on 8 participants recruited to Arm I. Adverse event reporting was not required, per protocol, for participants on Arm II (observation); therefore, there are no adverse event data to report for this arm.
Arm/Group | Arm II (Observation) | Arm I (Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/8
Other Adverse Events (participants affected / at risk) | 0/0 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Observation) (N=0) | Arm I (Chemotherapy) (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Observation) (N=0) | Arm I (Chemotherapy) (N=8)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (5)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (4)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less